CLINICAL TRIAL: NCT00004200
Title: A Randomized Double-Blind, Placebo-Controlled Phase II Study of the Matrix Metalloprotease Inhibitor Prinomastat in Combination With Temozolomide Following Radiation Therapy in Patients Having Newly Diagnosed Glioblastoma Multiforme
Brief Title: Prinomastat Plus Temozolomide Following Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AG-3340-019; CDR0000067443; MCC-12151; MDA-DM-99254; MSKCC-99116
Record Dates: First submitted 2000-01-21; First posted 2004-05-25 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — prinomastat; Temozolomide

INTERVENTIONS:
Drug: prinomastat
Drug: temozolomide

SUMMARY:
RATIONALE: Prinomastat may stop the growth of glioblastoma multiforme by stopping blood flow to the tumor. Drugs used in chemotherapy stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to study the effectiveness of prinomastat plus temozolomide in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the one year survival rate and progression free survival of patients with newly diagnosed glioblastoma multiforme treated with prinomastat (AG3340) or placebo and temozolomide following radiotherapy. II. Compare the safety of these regimens in these patients. III. Compare the quality of life in these patients on these regimens.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients receive oral prinomastat or placebo twice daily in combination with oral temozolomide daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed glioblastoma multiforme Must have completed all appropriate subtotal or total surgical procedures (surgical biopsy alone not eligible) Must have received prior external beam radiotherapy No multifocal glioblastoma multiforme No radiographic disease progression during post surgical radiotherapy

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Stable steroid therapy for at least 2 weeks prior to study Radiotherapy: See Disease Characteristics No prior interstitial brachytherapy or radiosurgery Surgery: See Disease Characteristics No prior radiosurgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Collier, Study Chair — Agouron Pharmaceuticals
Locations (1):
- Agouron Pharmaceuticals, Inc., La Jolla, California, United States